CLINICAL TRIAL: NCT04652895
Title: Sleep Quality, Heart Rate Variability and Anxiety Following Brain Injury
Status: Completed | Type: Observational
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, David Ripley, Principle Investigator, Shirley Ryan AbilityLab
Other Study IDs: STU00212891
Record Dates: First submitted 2020-10-16; First posted 2020-12-03 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Traumatic Brain Injury; Anxiety
Keywords: heart rate variability; sleep
MeSH Terms: conditions — Brain Injuries, Traumatic; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Moderate-to-severe traumatic brain injury inpatients: Moderate-to-severe traumatic brain injury inpatients

SUMMARY:
The investigators predict that decreased heart rate variability and poor sleep quality will be significantly correlated with higher self-reported anxiety following brain injury.

DETAILED DESCRIPTION:
Acute rehabilitation inpatients with moderate-to-severe brain injury will wear biosensors that track total sleep time and heart-rate variability for up to 1 week. During this time the participants will also complete surveys regarding symptoms of anxiety. The investigators hypothesize that decreased heart rate variability and poor sleep quality will be significantly correlated with higher self-reported anxiety following brain injury.

ELIGIBILITY:
Inclusion Criteria:

* traumatic brain injury
* injury within past 6 months
* medically stable
* able to communicate

Exclusion Criteria:

* on medication: beta-blocker
* adverse skin reaction to biosensor adhesive
* non-English speaking
* pregnant women
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: moderate to severe traumatic brain injury inpatients in acute rehabilitation hospital
Sampling Method: Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
anxiety | 48 hours
  self-reported anxiety survey

SECONDARY OUTCOMES:
heart rate variability | 48 hours
  Skin biosensor on patient chest, measuring heart rate over 6 minute interval while patient is awake and resting. Then heart rate variability is calculated based on the R-R interval.
sleep | 48 hours
  self-reported sleep survey. Also skin biosensor measuring heart rate and accelerometer overnight for 2 consecutive nights. Total sleep time and awakening episodes will be derived from the biosensor data.
post-traumatic stress disorder (PTSD) | 48 hours
  self-reported survey of PTSD symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Shirley Ryan Ability Lab, Chicago, Illinois, United States

DOCUMENTS (2):
  • Study Protocol (2020-08-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT04652895/Prot_000.pdf
  • Informed Consent Form (2020-09-11): https://cdn.clinicaltrials.gov/large-docs/95/NCT04652895/ICF_001.pdf